CLINICAL TRIAL: NCT06550726
Title: High-resolution Multi-parametric Magnetic Resonance Imaging for Focal Epilepsy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Leung Ho Sang, Associate Consultant, Department of Imaging and interventional Radiology, Prince of Wales Hospital, the Chinese University of Hong Kong, Chinese University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CREC 2024.133
Record Dates: First submitted 2024-08-05; First posted 2024-08-13 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Epilepsies, Partial
MeSH Terms: conditions — Epilepsies, Partial | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Masking Description: No masking is performed during the study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study subjects (Experimental): Study subjects will be recruited for scanning in a 3T MRI scanner with dedicated high-resolution MRI sequences as stated in our research protocol.
  Interventions: Diagnostic Test: Magnetic Resonance Imaging

INTERVENTIONS:
Diagnostic Test: Magnetic Resonance Imaging — Subjects will undergo MRI scanning in our 3T machine with dedicated high resolution sequences (including 2D T1-weighted inversion recovery sequences, 3D FLAIR MRI whole brain, 3D T1-weighted Sagittal MPRAGE; plus other sequences for the clinical purpose of pre-operative planning as per consensus with referring doctor)

SUMMARY:
Patients with focal epilepsy often have diagnostic difficulties as their culprit for seizures are difficult to be picked up using conventional imaging. The current study is to investigate the utility of advanced MRI sequences on detection of subtle lesions accountable for focal epilepsy.

DETAILED DESCRIPTION:
Focal epilepsy refers to having seizures arising from a specific part of the brain. In these patients, workup in magnetic resonance imaging is often necessary as patients with structural lesions have a much higher rate of seizures, ranging from 10% to 26% at 1 year and from 29% to 48% at 5 years. However, there is also a subgroup of patients who has epilepsy not adequately controlled by anti-epileptics with unrevealing first MRI study, a dedicated MRI protocol may reveal positive lesion in 30-65% of the cases. In these patients, several tricks can be applied to increase the detection rate. First, the used of a high-resolution MRI on a high-field scanner could be helpful, which can be increased the sensitivity up to 90%. The use of 7T-MRI in further picking up subtle lesions in patients presenting with epilepsy has been investigated, further affirming the role of high resolution MRI imaging. Secondly, the use of dedicated sequences, such as T1-weighted inversion recovery sequences which allow better distinction of grey and white matter, could also reveal subtle lesions such as polymicrogyria or Type 1 focal cortical dysplasia.

This study is therefore aimed to apply the findings to the local settings, and specifically to investigate if T1-weighted inversion recovery sequences provides additional benefit in picking up more subtle lesions in patients who had an initial first negative MRI.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive patients with drug-resistant focal epilepsy fulfilling the following criteria -

  1. Diagnosis of focal epilepsy with a probable site identified, as defined by concordant results from any TWO of the following:
* Clinical seminology compatible with focal epilepsy.
* Electroencephalography pointing towards a specific site for focal epilepsy.
* Positive ictal brain scintigraphy with SPECT-CT correlation. AND 2. Previous MRI (at least one study with protocol tailored for epilepsy) which did not reveal accountable focal lesion.

AND 3. Able to consent for MRI examination (if patient under age of 18, consent for MRI will be obtained from guardian). Patients will be provided information leaflets to read on, and written consent before taking part in this study and MRI examination.

Exclusion Criteria:

* Patients who are contraindicated to magnetic resonance imaging (such as due to underlying MRI incompatible metallic implants)
* Patients who cannot cooperate for MRI scanning.
* Patients show are unable to provide informed consent.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Accuracy of high resolution MRI in diagnosis | At the time of MRI scanning, typically 1 day
  the sensitivity and specificity of the baseline MRI (bMRI) and the high-resolution MRI (hrMRI) studies, based on the standard of surgical findings on patients who underwent either intracranial EEG or surgical resection

CONTACTS AND LOCATIONS:
Overall Officials: Hanson Leung, MBBS (HK), Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Gerald Choa MRI Center, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided
The image data and outcome measures of the participants can be provided in an anonymized manner upon reasonable request by email to the principal investigator.

REFERENCES:
- [Background] Scheffer IE, Berkovic S, Capovilla G, Connolly MB, French J, Guilhoto L, Hirsch E, Jain S, Mathern GW, Moshe SL, Nordli DR, Perucca E, Tomson T, Wiebe S, Zhang YH, Zuberi SM. ILAE classification of the epilepsies: Position paper of the ILAE Commission for Classification and Terminology. Epilepsia. 2017 Apr;58(4):512-521. doi: 10.1111/epi.13709. Epub 2017 Mar 8. PMID 28276062
- [Background] Bernasconi A, Cendes F, Theodore WH, Gill RS, Koepp MJ, Hogan RE, Jackson GD, Federico P, Labate A, Vaudano AE, Blumcke I, Ryvlin P, Bernasconi N. Recommendations for the use of structural magnetic resonance imaging in the care of patients with epilepsy: A consensus report from the International League Against Epilepsy Neuroimaging Task Force. Epilepsia. 2019 Jun;60(6):1054-1068. doi: 10.1111/epi.15612. Epub 2019 May 28. PMID 31135062
- [Background] Krumholz A, Wiebe S, Gronseth GS, Gloss DS, Sanchez AM, Kabir AA, Liferidge AT, Martello JP, Kanner AM, Shinnar S, Hopp JL, French JA. Evidence-based guideline: Management of an unprovoked first seizure in adults: Report of the Guideline Development Subcommittee of the American Academy of Neurology and the American Epilepsy Society. Neurology. 2015 Apr 21;84(16):1705-13. doi: 10.1212/WNL.0000000000001487. PMID 25901057
- [Background] Kokkinos V, Kallifatidis A, Kapsalaki EZ, Papanikolaou N, Garganis K. Thin isotropic FLAIR MR images at 1.5T increase the yield of focal cortical dysplasia transmantle sign detection in frontal lobe epilepsy. Epilepsy Res. 2017 May;132:1-7. doi: 10.1016/j.eplepsyres.2017.02.018. Epub 2017 Mar 2. PMID 28279892
- [Background] Mellerio C, Labeyrie MA, Chassoux F, Roca P, Alami O, Plat M, Naggara O, Devaux B, Meder JF, Oppenheim C. 3T MRI improves the detection of transmantle sign in type 2 focal cortical dysplasia. Epilepsia. 2014 Jan;55(1):117-22. doi: 10.1111/epi.12464. Epub 2013 Nov 15. PMID 24237393
- [Background] Hou P, Hasan KM, Sitton CW, Wolinsky JS, Narayana PA. Phase-sensitive T1 inversion recovery imaging: a time-efficient interleaved technique for improved tissue contrast in neuroimaging. AJNR Am J Neuroradiol. 2005 Jun-Jul;26(6):1432-8. PMID 15956512

DOCUMENTS (2):
  • Study Protocol (2024-04-18): https://cdn.clinicaltrials.gov/large-docs/26/NCT06550726/Prot_000.pdf
  • Informed Consent Form (2024-04-18): https://cdn.clinicaltrials.gov/large-docs/26/NCT06550726/ICF_001.pdf